CLINICAL TRIAL: NCT04421378
Title: A Phase 1/2 Study of Selinexor in Combination With Standard of Care (SoC) Therapy for Newly Diagnosed or Recurrent Glioblastoma
Brief Title: A Study of Selinexor in Combination With Standard of Care Therapy for Newly Diagnosed or Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Upon further consideration of the existing data and the competitive landscape, Karyopharm Therapeutics Inc has decided not to pursue the ongoing development of Selinexor in GBM at this time.
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-GBM-029; 2021-000080-67 (EudraCT Number)
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma Multiforme
Keywords: nGBM; rGBM; GBM; Temozolomide; Lomustine; KPT-330; XPOVIO; Selinexor; Newly diagnosed glioblastoma multiforme; Recurrent glioblastoma multiforme; Bevacizumab; TTField
MeSH Terms: conditions — Glioblastoma | interventions — selinexor; Temozolomide; Lomustine; Bevacizumab; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1: Arm A: Selinexor+Radiation Therapy (Experimental): Participants with nGBM uMGMT will receive 60 to 80 milligram (mg) of selinexor oral tablet once weekly (QW) across dose level -1, 1, 2, and 3 in combination with 2 Gray (Gy) radiation therapy (RT) daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 80 mg of selinexor oral tablet on Day 1 and 15 in a 28-day Cycle 2 and subsequently will continue at 80 mg QW until progressive disease (PD) during adjuvant therapy period.
  Interventions: Drug: Selinexor; Radiation: Standard Fractionated Radiation therapy (RT)
- Arm A Control: Temozolomide+Radiation Therapy (Active Comparator): Participants with nGBM uMGMT will receive 75 milligram per meter square (mg/m^2) of temozolomide oral capsule once daily (QD) in combination with 2 Gy RT daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 150 mg/m^2 (started from Cycle 3) and increase to 200 mg/m^2 as tolerated per Investigator's judgment, daily for 5 days in a 28-day cycle during Cycles 4 to 8 cycles during adjuvant therapy period.
  Interventions: Drug: Temozolomide (TMZ); Radiation: Standard Fractionated Radiation therapy (RT)
- Phase 1: Arm B: Selinexor+Temozolomide+Radiation Therapy (Experimental): Participants with nGBM mMGMT will receive 40-80 mg of selinexor oral tablet QW across dose level -1, 1, 2, 2a, 2b and 3a and 75 mg/m^2 of temozolomide oral capsule QD in combination with 2 Gy RT daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 60 mg (dose level 2a) or 80 mg (dose level 2b and 3a) of selinexor oral tablet on Day 1 and 15 in a 28-day Cycle 2, followed by 150 mg/m^2 (started from Cycle 3) and increase to 200 mg/m^2 as tolerated per Investigator's judgment, daily for 5 days in a 28-day cycle during Cycle 4 to 8 during adjuvant therapy period. Participants will continue selinexor weekly per dose level assigned until PD.
  Interventions: Drug: Selinexor; Drug: Temozolomide (TMZ); Radiation: Standard Fractionated Radiation therapy (RT)
- Arm B Control: Temozolomide+Radiation Therapy (Active Comparator): Participants with nGBM mMGMT will receive 75 mg/m^2 of temozolomide oral capsule QD in combination with 2 Gy RT daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 150 mg/m^2 (started from Cycle 3) and increase to 200 mg/m^2 as tolerated per Investigator's judgment, daily for 5 days in a 28-day cycle during Cycles 4 to 8 during adjuvant therapy period.
  Interventions: Drug: Temozolomide (TMZ); Radiation: Standard Fractionated Radiation therapy (RT)
- Arm C: Selinexor+Lomustine/Carmustine (Experimental): Participants with rGBM uMGMT or mMGMT will receive 40-80 mg of selinexor oral tablet QW across dose level -1, 1, 2, 2a, and 3 and 90-110 mg/m^2 of lomustine or 150-200 mg/m^2 of carmustine (substituted if lomustine is not available) capsule on Day 1 of each cycle across dose level -1, 1, 2, 2a, and 3 in a 42-day cycle for all cycles.
  Interventions: Drug: Selinexor; Drug: Lomustine (CCNU); Drug: Carmustine
- Arm C Control: Lomustine/Carmustine (Active Comparator): Participants with rGBM uMGMT or mMGMT will receive 110 mg/m^2 of lomustine or 200 mg/m^2 of Carmustine (substituted if lomustine is not available) capsule on Day 1 of each cycle in a 42-day cycle for all cycles.
  Interventions: Drug: Lomustine (CCNU); Drug: Carmustine
- Arm D: Selinexor+Bevacizumab (Experimental): Participants with rGBM will receive 60-80 mg of selinexor oral tablet QW across dose level -1, 1 and 10 mg/kg of Bevacizumab intravenous (IV) infusion every 2 weeks (Q2W) in 28-day cycle for all cycles.
  Interventions: Drug: Selinexor; Drug: Bevacizumab
- Arm E: Selinexor+TTField (Experimental): Participants with rGBM will receive 60-80 mg of selinexor oral tablet QW across dose level -1, 1 and will receive scalp application of 200 kilohertz (kHz) of transducer array ≥18 hours/day daily for each cycle in 28 day cycle for all cycles.
  Interventions: Drug: Selinexor; Device: TTField

INTERVENTIONS:
Drug: Selinexor — Dose and Formulation: 20 milligram (mg); Tablet Route of Administration: Oral
  Other Names: KPT-330; XPOVIO
  Arms: Arm C: Selinexor+Lomustine/Carmustine; Arm D: Selinexor+Bevacizumab; Arm E: Selinexor+TTField; Phase 1: Arm A: Selinexor+Radiation Therapy; Phase 1: Arm B: Selinexor+Temozolomide+Radiation Therapy
Drug: Temozolomide (TMZ) — Dose strength and Formulation: 5, 20, 100, 140, 180, or 250 mg; Capsule Route of Administration: Oral
  Other Names: Temodar
  Arms: Arm A Control: Temozolomide+Radiation Therapy; Arm B Control: Temozolomide+Radiation Therapy; Phase 1: Arm B: Selinexor+Temozolomide+Radiation Therapy
Drug: Lomustine (CCNU) — Dose and Formulation: 10, 40, or 100 mg; Capsule Route of Administration: Oral
  Arms: Arm C Control: Lomustine/Carmustine; Arm C: Selinexor+Lomustine/Carmustine
Radiation: Standard Fractionated Radiation therapy (RT) — Radiation Therapy Oncology Group (RTOG) or European Organisation for Research and Treatment of Cancer (EORTC) methodologies of approximately 60 Gy in 30 fractions.
  Arms: Arm A Control: Temozolomide+Radiation Therapy; Arm B Control: Temozolomide+Radiation Therapy; Phase 1: Arm A: Selinexor+Radiation Therapy; Phase 1: Arm B: Selinexor+Temozolomide+Radiation Therapy
Drug: Bevacizumab — Dose and Formulation: 10 mg/kg; Route of Administration: Intravenous
  Arms: Arm D: Selinexor+Bevacizumab
Device: TTField — Dose and Formulation: 200 kHz ≥18h/day; Route of administration: Scalp application of transducer arrays.
  Arms: Arm E: Selinexor+TTField
Drug: Carmustine — Dose and Formulation: 150 or 200 mg/m^2; Route of Administration: Intravenous
  Arms: Arm C Control: Lomustine/Carmustine; Arm C: Selinexor+Lomustine/Carmustine

SUMMARY:
This is a Phase 1/2 study of selinexor in combination with standard of care (SoC) therapy for newly diagnosed glioblastoma (nGBM) or recurrent glioblastoma (rGBM). This study will be conducted in 2 phases: a Phase 1a dose finding study followed by Phase 1b (dose expansion) and a Phase 2 randomized efficacy exploration study and will independently evaluate 3 different combination regimens in 3 treatment arms in patients with nGBM (Arms A and B) or with rGBM (Arm C).

* Arm A: evaluating the combination of selinexor with radiation therapy (S-RT) in nGBM participants with uMGMT
* Arm B: evaluating the combination of selinexor with radiation therapy and temozolomide (TMZ) (S-TRT) in nGBM participants with methylated-O6-methylguanine-DNA-methyltransferase (mMGMT)
* Arm C: evaluating the combination of selinexor with lomustine (or carmustine, if lomustine is not available) (S-L/C) in rGBM participants regardless of MGMT status
* Arm D: evaluating the combination of selinexor with bevacizumab in rGBM participants regardless of MGMT status
* Arm E: evaluating the combination of selinexor with tumor treating fields (TTField) in rGBM participants regardless of MGMT status

ELIGIBILITY:
Inclusion Criteria

* Written informed consent in accordance with federal, local, and institutional guidelines.
* Age ≥18 years at the time of informed consent and ≥22 year for Arm E.
* Pathologically confirmed glioblastoma (including all histological variants; documentation to be provided) that are newly diagnosed (for Arms A and B) or relapsed disease (for Arm C, D and E) after 1 to 2 line of systemic therapy (RT ± TMZ or RT ± TMZ in combination with other drug) (surgical resection of recurrent disease allowed). For Arms A and B, MGMT status should be available.
* Prior therapy:

  1. Arms A and B: participants who have not received RT or any systemic therapy for brain tumor and must be eligible for definitive external beam RT and TMZ
  2. Arm C, D and E: participants must have received prior treatment with RT with or without TMZ and only 1 prior line of therapy (RT ± TMZ in combination with other drug is allowed).
* Measurable disease according to RANO/modified RANO guidelines is required only for Arm C, D and E; it is not required for Arms A or B.
* Participants enrolling into Arms C, D, and E must be on a stable or decreasing dose of corticosteroids (or none) for at least 5 days prior to the baseline magnetic resonance imaging (MRI).
* Karnofsky Performance Score (KPS) ≥70 (for Arms A and B) and 60 (for Arms C, D, and E).
* Participants must have adequate organ function ≤2 weeks of study treatment as defined by the following laboratory criteria:

  1. Hematological function ≤7 days prior to Cycle 1 Day 1 (C1 D1): Absolute neutrophil count (ANC) ≥1.5*10^9 per Liter (/L); platelet count ≥150*10^9/L; and hemoglobin (Hb) ≥10.0 gram per deciliter (g/dL). Transfusion is not allowed within 7 days prior to C1 D1
  2. Hepatic function: bilirubin ≤2*the upper limit of normal (ULN), alanine transaminase (ALT) ≤2.5*ULN, aspartate transaminase (AST) ≤2.5*ULN; unless bilirubin elevation is related to Gilbert's Syndrome for which bilirubin must be <4*ULN
  3. Renal function: calculated (Cockcroft-Gault) or measured creatinine clearance ≥30 milliliter per minute (mL/min)
* Female participants of childbearing potential must have a negative serum pregnancy test at Screening and agree to use highly effective methods of contraception throughout the study and for 6 months following the last dose of study treatment.
* Fertile male participants who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 6 months following the last dose of study treatment.
* For Arms A and B: participants must have had surgery and/or biopsy not greater than [>] 8 weeks prior to initial screening.
* Participants must consent to provide tumor tissue and blood samples to be used for future molecular testing for correlative studies.
* Limited to supratentorial disease for Arm E only.

Exclusion Criteria

- Participants who are receiving any other investigational agents and /or have had prior therapy including:

For Arms A and B only:

1. Participants who have previously received RT to the brain
2. Participants who received chemotherapy for the treatment of their glioma
3. Participants who are being treated with implanted Gliadel wafers

   For Arm C:
4. Prior nitrosoureas

   For Arms C, D, and E:
5. <4 weeks from prior TMZ or other chemotherapy, or <4 weeks or 5 half-lives (whichever is shorter) for investigational agents prior to start of study treatment
6. Prior treatment bevacizumab or other direct Vascular endothelial growth factor/Vascular endothelial growth factor receptor (VEGF/VEGFR) inhibitors. For any questions of the definition of a direct VEGF/VEGFR inhibitor, consult the study Medical Monitor
7. Any AE which has not recovered to Grade <=1, or returned to baseline, related to the previous GBM therapy, except alopecia, and some other Grade 2 AEs that have been stabilized (upon Medical Monitor approval)

   * Participants who are being treated or plan to be treated during this study with TTField for participants in Arms A to D.
   * Major surgery <2 weeks prior to the start of study treatment for Arms A to C and E, <4 weeks for Arm D.
   * History of allergic reactions attributed to compounds of similar chemical or biological composition to selinexor or other study treatment.
   * Participants must not have significantly diseased or obstructed gastrointestinal tract malabsorption, uncontrolled vomiting or diarrhea, or inability to swallow oral medication.
   * Participants with coagulation problems and medically significant bleeding in the month prior to start of treatment (peptic ulcers, epistaxis, intracranial hemorrhage, spontaneous bleeding). Prior history of deep vein thrombosis or pulmonary embolism is not exclusionary.
   * Currently pregnant or breastfeeding.
   * For Arms A and B: participants with pre-existing known or suspected radiation sensitivity syndromes will be excluded due to potential confounding effect on outcome.
   * Any life-threatening illness, active medical condition, organ system dysfunction, or serious active psychiatric issue which, in the Investigator's opinion, could compromise the participant's safety or the participant's ability to remain compliant with study procedures.
   * Uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within 7 days prior to first dose of study treatment; however, prophylactic use of these agents is acceptable even if parenteral.
   * Participants with mutated isocitrate dehydrogenase (IDH) should be excluded for Phase 2.
   * For participants in Arm C, Forced Vital Capacity (FVC) or Carbon Monoxide Diffusing Capacity (DLCO) below 70% of predicted.
   * For Arm E: implanted active electronic medical devices such as programmable intraventricular shunts, spinal cord, vagus nerve or deep brain stimulators, pacemakers or implantable automatic defibrillators, skull defect (i.e. missing bone with no replacement), sensitivity to conductive hydrogels as used in electrocardiograms (ECGs), an underlying serious scalp condition that may interfere with placement of arrays, or bullet fragments, or documented clinically significant arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Lassman, MD, Principal Investigator — Columbia University
Locations (18):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - University of Southern California (USC Norris Comprehensive Cancer Center and LAC+USC Medical Center), Los Angeles, California
  - University of California, San Francisco, California
  - Baptist Hospital of Miami Cancer Institute, 8900 North Kendall Drive, Miami, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack Meridian Health, 92 Second Street, Hackensack, New Jersey
  - Atlantic Health Systems Hospital Corp., Morristown, New Jersey
  - Northwell Health, Lake Success, New York
  - Columbia University Irving Medical Center, New York, New York
  - Lenox Hill Hospital-Northwell Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington - Alvord Brain Tumor Center, Seattle, Washington
- Princess Margaret Hospital (PMH), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 18 sites in the United States and Canada. This study had three phases: Phase 1a, Phase 1b and Phase 2. The study was early terminated during the Phase 1b portion of the study as the initial responses to selinexor treatment were not supportive of continued investigation in glioblastoma, therefore Phase 2 data could not be collected and there was no reporting of the Phase 2 data in this report.
Pre-assignment Details: Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Groups:
- Arm A: Selinexor + Radiation Therapy: Participants with newly diagnosed glioblastoma (nGBM) unmethylated O6-methylguanine-DNA-methyltransferase (uMGMT) received 60 to 80 milligrams (mg) of selinexor oral tablet, once weekly (QW) in combination with 2 Gray (Gy) radiation therapy (RT) daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 80 mg of selinexor oral tablet on Day 1 and 15 in a 28-day Cycle 2 and subsequently continued at 80 mg of selinexor, QW until progressive disease (PD) during adjuvant therapy period.
- Arm B: Selinexor + Temozolomide + Radiation Therapy: Participants with nGBM methylated O6-methylguanine-DNA-methyltransferase (mMGMT) received 40 to 80 mg of selinexor oral tablet, QW and 75 milligrams per sqaure meter (mg/m^2) of temozolomide oral capsule, once daily (QD) in combination with 2 Gy RT daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 60 mg or 80 mg of selinexor oral tablet on Day 1 and 15 in a 28-day Cycle 2, followed by 150 mg/m^2 of temozolomide oral capsule and increase to 200 mg/m^2, daily for 5 days in a 28-day cycle during Cycle 3 to 8 during adjuvant therapy period. Participants continued selinexor weekly until PD.
- Arm C: Selinexor + Lomustine/Carmustine: Participants with recurrent glioblastoma (rGBM) uMGMT or mMGMT received 40 to 80 mg of selinexor oral tablet, QW and 90 to 110 mg/m^2 of lomustine or 150 to 200 mg/m^2 of carmustine (substituted if lomustine is not available) capsule on Day 1 of each 42-days cycle for up to 6 cycles. Participants continued selinexor weekly until PD.
- Arm D: Selinexor + Bevacizumab: Participants with rGBM received 60 to 80 mg of selinexor oral tablet, QW and 10 mg/kg of Bevacizumab intravenous (IV), infusion every 2 weeks (Q2W) in each 28-day cycle until PD, unacceptable adverse events (AEs) or failure to tolerate the study treatment, treatment delay of more than 28 days (except in specific cases with documented approval from the Sponsor), any medically appropriate reason or significant protocol violation (in the opinion of the Investigator), or participant decided to discontinue study treatment, withdraws consent, or became pregnant.
- Arm E: Selinexor + Tumor Treating Fields: Participants with rGBM received 60 to 80 mg of selinexor oral tablet, QW and received scalp application of 200 kilohertz (kHz) of transducer array greater than or equal to (>=) 18 hours per day daily for each 28-day cycle until PD, unacceptable AEs or failure to tolerate the study treatment, treatment delay of more than 28 days (except in specific cases with documented approval from the Sponsor), any medically appropriate reason or significant protocol violation (in the opinion of the Investigator), or participant decided to discontinue study treatment, withdraws consent, or became pregnant.
Period: Overall Study
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Started | 23 | 15 | 19 | 14 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 15 | 19 | 14 | 3
Not completed — Adverse Event | 2 | 7 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 16 | 4 | 18 | 11 | 3
Not completed — Study Terminated by Sponsor | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 2 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of participants who have been assigned to study intervention and who have received >=1 dose of study drug. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Groups:
- Arm A: Selinexor + Radiation Therapy: Participants with nGBM uMGMT received 60 to 80 mg of selinexor oral tablet, once QW in combination with 2 Gy RT daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 80 mg of selinexor oral tablet on Day 1 and 15 in a 28-day Cycle 2 and subsequently continued at 80 mg of selinexor, QW until PD during adjuvant therapy period.
- Arm B: Selinexor + Temozolomide + Radiation Therapy: Participants with nGBM mMGMT received 40 to 80 mg of selinexor oral tablet, QW and 75 mg/m^2 of temozolomide oral capsule, QD in combination with 2 Gy RT daily for 5 days per week in a 42-day cycle during Cycle 1 radiation period followed by 60 mg or 80 mg of selinexor oral tablet on Day 1 and 15 in a 28-day Cycle 2, followed by 150 mg/m^2 of temozolomide oral capsule and increase to 200 mg/m^2, daily for 5 days in a 28-day cycle during Cycle 3 to 8 during adjuvant therapy period. Participants continued selinexor weekly until PD.
- Arm C: Selinexor + Lomustine/Carmustine: Participants with rGBM uMGMT or mMGMT received 40 to 80 mg of selinexor oral tablet, QW and 90 to 110 mg/m^2 of lomustine or 150 to 200 mg/m^2 of carmustine (substituted if lomustine is not available) capsule on Day 1 of each 42-days cycle for up to 6 cycles. Participants continued selinexor weekly until PD.
- Arm D: Selinexor + Bevacizumab: Participants with rGBM received 60 to 80 mg of selinexor oral tablet, QW and 10 mg/kg of Bevacizumab IV, infusion Q2W in each 28-day cycle until PD, unacceptable AEs or failure to tolerate the study treatment, treatment delay of more than 28 days (except in specific cases with documented approval from the Sponsor), any medically appropriate reason or significant protocol violation (in the opinion of the Investigator), or participant decided to discontinue study treatment, withdraws consent, or became pregnant.
- Arm E: Selinexor + Tumor Treating Fields: Participants with rGBM received 60 to 80 mg of selinexor oral tablet, QW and received scalp application of 200 kHz of transducer array >=18 hours per day daily for each 28-day cycle until PD, unacceptable AEs or failure to tolerate the study treatment, treatment delay of more than 28 days (except in specific cases with documented approval from the Sponsor), any medically appropriate reason or significant protocol violation (in the opinion of the Investigator), or participant decided to discontinue study treatment, withdraws consent, or became pregnant.
- Total: Total of all reporting groups
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields | Total
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.84) | 53.3 (14.88) | 59.2 (10.22) | 59.0 (10.50) | 53.3 (2.52) | 57.7 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 9 | 4 | 1 | 32
  Male | 12 | 8 | 10 | 10 | 2 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 1 | 4 | 1 | 14
  Not Hispanic or Latino | 17 | 13 | 17 | 10 | 2 | 59
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 1 | 0 | 4
  White | 23 | 12 | 16 | 13 | 3 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a and 1b: Maximum Tolerated Dose of Selinexor
Description: MTD was defined as highest dose of selinexor in at which no more than one of six participants experienced a dose-limiting toxicity (DLT). DLT was based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: At Cycle 1 (up to 42 days)
Population: The dose escalation population consisted of all participants in the Dose Escalation Phase who have either had a DLT prior to completion of 1 cycle of therapy, or who had completed a cycle of therapy. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Measure: Number; unit: milligrams per week
Groups:
- Arms A+B+C+D+E: Selinexor: All participants who received 40 to 80 mg or 60 to 80 mg of selinexor oral tablet, QW in each 28-day cycle until PD.
Arm/Group | Arms A+B+C+D+E: Selinexor
Number analyzed (Participants) | 74
milligrams per week | 60

2. Primary Outcome: Phase 1a and 1b: Recommended Phase 2 Dose (RP2D) of Selinexor
Description: The RP2D was determined by SRC, based on the MTD and the totality of efficacy and safety data of Phase 1a dose escalation study. RP2D was determined based on the totality of the available safety, efficacy, pharmacokinetic/pharmacodynamic (PK/PD).
Time Frame: From Cycle 1 Day 1 up to 14 days after last dose (up to 15.41 months) (Each Cycle length = up to 42 days)
Population: as for outcome 1
Measure: Number; unit: milligrams per week
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3
milligrams per week | 80 | NA — Here 'NA' means RP2D could not be determined as Arm B was still in dose finding when the study terminated. | NA — Here 'NA' means RP2D could not be determined as Arm C was still in dose finding when the study terminated. | 80 | NA — Here 'NA' means RP2D could not be determined as the number of participants was considered too small for any definitive conclusions.

3. Primary Outcome: Phase 1a and 1b: Number of Participants With Treatment-emergent Adverse Events (TEAEs) With Grade Greater Than or Equal to (>=) 3, Serious TEAEs and Who Discontinued Treatment Due to TEAEs
Description: TEAE: any event that was not present prior to initiation of study treatment or any event already present that worsened in either intensity or frequency following exposure to study treatment. Serious adverse event (SAE): any untoward medical occurrence that, at any dose, resulted in death; was life threatening (i.e., an event in which participant was at risk of death at the time of the event; it did not refer to an event that hypothetically might have caused death if it were more severe); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; or was a congenital anomaly/birth defect. Important medical events that might not result in death, was life-threatening, or require hospitalization might be considered serious when, based upon appropriate medical judgment, they might jeopardize participant and might require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From first dose of study treatment up to 30 days post last dose (Up to 16.41 months)
Population: The safety population consisted of participants in Phase 1a and Phase 1b who have been assigned to study intervention and who have received >=1 dose of study drug. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3
Participants
  Participants with Grade >=3 TEAEs | 15 | 12 | 16 | 8 | 1
  Participants with Serious TEAEs | 6 | 5 | 6 | 3 | 1
  Participants who Discontinued Treatment Due to TEAEs | 2 | 7 | 0 | 1 | 0

4. Primary Outcome: Phase 1a and 1b: Percentage of Participants With Progression Free Survival at 3 Months
Description: Progression defined as first occurrence of disease progression (PD) per modified Response Assessment in Neuro-Oncology (RANO) including both radiological PD and clinical deterioration. PD per RANO response criteria:1) At least two sequential scans separated by at >=4 weeks both exhibiting >=25 percent (%) increase in sum of products of perpendicular diameters or >=40% increase in total volume of enhancing lesions. 2) In case where baseline or best response demonstrates no measurable enhancing disease, then any new measurable (>10mm*10mm) enhancing lesions considered PD after confirmed by a subsequent scan >=4 weeks exhibiting >=25% increase in sum of products of perpendicular diameters or >=40% increase in total volume of enhancing lesions relative to scan first illustrating new measurable disease. 3) Clear clinical deterioration not attributable to other causes apart from tumor or attributable to changes in steroid dose. 4) Failure to return for evaluation as a result of death.
Time Frame: At 3 Months
Population: The modified Intent-to-Treat (mITT) population consisted of participants in Phase 1a and Phase 1b who have been assigned to study intervention and who have received >=1 dose of study drug. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3
percentage of participants | 69.6 | 66.7 | 21.1 | 57.1 | 33.3

5. Primary Outcome: Phase 1a and 1b: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until death due to any cause or until lost to follow-up for all participants.
Time Frame: From date of randomization to the date of death due to any cause or until lost to follow-up (up to 20 months)
Population: The mITT population consisted of participants in Phase 1a and Phase 1b who have been assigned to study intervention and who have received >=1 dose of study drug. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3
months | 13.54 [11.37 to 18.23] | 19.78 [13.50 to NA] — Here, NA means data could not be determined due to insufficient events. | 8.34 [7.13 to 12.75] | 8.80 [6.05 to NA] — Here, NA means data could not be determined due to insufficient events. | 14.36 [7.20 to NA] — Here, NA means data could not be determined due to insufficient events.

6. Secondary Outcome: Phase 1a and 1b: Time to Progression (TTP)
Description: TTP was defined for participants as the duration from start of treatment to the date of PD, or death due to PD, whichever occurs first. PD per RANO response criteria: 1) At least two sequential scans separated by at >=4 weeks both exhibiting >=25 percent (%) increase in sum of products of perpendicular diameters or >=40% increase in total volume of enhancing lesions. 2) In case where baseline or best response demonstrates no measurable enhancing disease, then any new measurable (>10mm*10mm) enhancing lesions considered PD after confirmed by a subsequent scan >=4 weeks exhibiting >=25% increase in sum of products of perpendicular diameters or >=40% increase in total volume of enhancing lesions relative to scan first illustrating new measurable disease. 3) Clear clinical deterioration not attributable to other causes apart from tumor or attributable to changes in steroid dose. 4) Failure to return for evaluation as a result of death or deteriorating condition.
Time Frame: From first dose study treatment until progression or death due to progression (Up to 15.41 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3
months | 8.11 [6.05 to 11.50] | NA [11.37 to NA] — Here, NA means data could not be determined due to insufficient events. | 1.38 [1.22 to 4.07] | 4.60 [2.53 to NA] — Here, NA means data could not be determined due to insufficient events. | 1.71 [1.64 to NA] — Here, NA means data could not be determined due to insufficient events.

7. Secondary Outcome: Phase 1a and 1b: Progressive Free Survival (PFS)
Description: Progression defined as first occurrence of PD per modified RANO including both radiological PD and clinical deterioration. PD per RANO response criteria: 1) At least two sequential scans separated by at >=4 weeks both exhibiting >=25 percent (%) increase in sum of products of perpendicular diameters or >=40% increase in total volume of enhancing lesions. 2) In case where baseline or best response demonstrates no measurable enhancing disease, then any new measurable (>10mm*10mm) enhancing lesions considered PD after confirmed by a subsequent scan >=4 weeks exhibiting >=25% increase in sum of products of perpendicular diameters or >=40% increase in total volume of enhancing lesions relative to scan first illustrating new measurable disease. 3) Clear clinical deterioration not attributable to other causes apart from tumor or attributable to changes in steroid dose. 4) Failure to return for evaluation as a result of death or deteriorating condition.
Time Frame: From first dose of study treatment until progression or death due to any cause (Up to 15.41 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 23 | 15 | 19 | 14 | 3
months | 8.11 [6.05 to 11.50] | NA [11.37 to NA] — Here, NA means data could not be determined due to insufficient events. | 1.38 [1.22 to 4.07] | 4.60 [2.53 to NA] — Here, NA means data could not be determined due to insufficient events. | 1.71 [1.64 to NA] — Here, NA means data could not be determined due to insufficient events.

8. Secondary Outcome: Phase 1a and 1b: Overall Response Rate (ORR) Based on Modified Response Assessment in Neuro-Oncology (RANO) Criteria in Arm C, D and E
Description: ORR was defined as percentage of participants who achieve a CR or PR per modified RANO criteria. CR defined as that meet all following: 1) Disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks. 2) No new lesions. 3) Participants must be off corticosteroids (or on physiologic replacement doses only). 4) Stable or improved clinical assessments (i.e., neurological examinations). PR defined as that meet all following: 1) >=50% decrease in sum of products of perpendicular diameters or >=65% decrease in total volume of all measurable enhancing lesions compared with baseline, sustained for at least 4 weeks. 2) No new lesion. 3. Steroid dose should be the same or lower compared with baseline scan. 4) Stable or improved clinical assessments.
Time Frame: From first dose of study treatment until death due to any cause (Up to 15.41 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 19 | 14 | 3
percentage of participants | 10.5 [1.3 to 33.1] | 35.7 [12.8 to 64.9] | 0 [NA to NA] — Here, NA means data could not be determined due to insufficient events.

9. Secondary Outcome: Phase 1a and 1b: Disease Control Rate (DCR) Based on Modified Response Assessment in Neuro-Oncology (RANO) Criteria in Arm C, D and E
Description: DCR: percentage of participants who achieve CR, PR, or stable disease (SD) per modified RANO criteria. CR: 1) Disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks. 2) No new lesions. 3) Participants must be off corticosteroids. 4) Stable or improved clinical assessments. PR: 1) >=50% decrease in sum of products of perpendicular diameters or >=65% decrease in total volume of all measurable enhancing lesions compared with baseline, sustained for at least 4 weeks. 2) No new lesion. 3) Steroid dose should be same or lower compared with baseline scan. 4) Stable or improved clinical assessments. SD: 1) Does not qualify for CR, PR, or PD. 2) In event that corticosteroid dose was increased without confirmation of PD on neuroimaging, and subsequent follow-up imaging shows steroid increase was required because of PD, last scan considered to show SD was scan obtained when corticosteroid dose was equivalent to baseline dose.
Time Frame: From first dose of study treatment until death due to any cause (Up to 15.41 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 19 | 14 | 3
percentage of participants | 21.1 [6.1 to 45.6] | 57.1 [28.9 to 82.3] | 0 [NA to NA] — Here, NA means data could not be determined due to insufficient events.

10. Secondary Outcome: Phase 1a and 1b: Duration of Response (DOR) in Arm C, D and E
Description: DOR was defined as the time from the date of first evidence of objective response (CR or PR) until PD. CR defined as that meet all following: 1) Disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks. 2) No new lesions. 3) Participants must be off corticosteroids (or on physiologic replacement doses only). 4) Stable or improved clinical assessments (i.e., neurological examinations). PR defined as that meet all following: 1) >=50% decrease in sum of products of perpendicular diameters or >=65% decrease in total volume of all measurable enhancing lesions compared with baseline, sustained for at least 4 weeks. 2) No new lesion. 3. Steroid dose should be the same or lower compared with baseline scan. 4) Stable or improved clinical assessments. DOR was analyzed by Kaplan-Meier for participants who have achieved overall response (CR or PR).
Time Frame: From the date of first evidence of objective response until progression (Up to 15.41 months)
Population: The mITT population. Here, "overall number of participants analyzed" signifies those participants who had CR or PR. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
Number analyzed (Participants) | 2 | 5 | 0
months | NA [3.02 to NA] — Here, NA means data could not be determined due to insufficient events. | 3.52 [2.79 to NA] — Here, NA means data could not be determined due to insufficient events. |

11. Secondary Outcome: Phase 1a and 1b: Maximum Plasma Concentration (Cmax) of Selinexor
Description: Cmax of Selinexor was reported.
Time Frame: Cycle 1 Day 1: 2, 4, and 6 hours post-dose (Cycle 1 length = up to 42 days)
Population: PK analysis set. Here, "overall number of participants analyzed" signifies those participants who are evaluable for this outcome. Due to the early study termination and pre-specified analysis, data was collected/reported for Cmax was calculated across treatment for each patient per dose level (40 mg, 60 mg and 80 mg) considering no accumulation of selinexor.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Selinexor 40 mg: Participants received 40 mg of selinexor oral tablet, once QW until PD.
- Selinexor 60 mg: Participants received 60 mg of selinexor oral tablet, once QW until PD.
- Selinexor 80 mg: Participants received 80 mg of selinexor oral tablet, once QW until PD.
Arm/Group | Selinexor 40 mg | Selinexor 60 mg | Selinexor 80 mg
Number analyzed (Participants) | 3 | 5 | 23
nanograms per milliliter (ng/mL) | 306 (17.8) | 490 (35.9) | 607 (32.3)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 30 days post last dose (Up to 20 months)
Description: The safety population consisted of participants who have been assigned to study intervention and who have received >=1 dose of study drug. Due to the early study termination and pre-specified analysis, data was collected/reported according to disease characteristics and combined dose range (60 to 80 mg or 40 to 80 mg) participants received regardless of study phase. The 'per arm' or 'per dose level' data was not collected.
Arm/Group | Arm A: Selinexor + Radiation Therapy | Arm B: Selinexor + Temozolomide + Radiation Therapy | Arm C: Selinexor + Lomustine/Carmustine | Arm D: Selinexor + Bevacizumab | Arm E: Selinexor + Tumor Treating Fields
All-Cause Mortality (participants affected / at risk) | 15/23 | 7/15 | 15/19 | 11/14 | 3/3
Serious Adverse Events (participants affected / at risk) | 6/23 | 5/15 | 6/19 | 3/14 | 1/3
Other Adverse Events (participants affected / at risk) | 23/23 | 15/15 | 19/19 | 14/14 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Selinexor + Radiation Therapy (N=23) | Arm B: Selinexor + Temozolomide + Radiation Therapy (N=15) | Arm C: Selinexor + Lomustine/Carmustine (N=19) | Arm D: Selinexor + Bevacizumab (N=14) | Arm E: Selinexor + Tumor Treating Fields (N=3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Agitation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Selinexor + Radiation Therapy (N=23) | Arm B: Selinexor + Temozolomide + Radiation Therapy (N=15) | Arm C: Selinexor + Lomustine/Carmustine (N=19) | Arm D: Selinexor + Bevacizumab (N=14) | Arm E: Selinexor + Tumor Treating Fields (N=3)
Neutropenia (Blood and lymphatic system disorders) | 12 | 11 | 11 | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 10 | 15 | 7 | 1
Lymphopenia (Blood and lymphatic system disorders) | 8 | 9 | 10 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 8 | 5 | 8 | 8 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 6 | 7 | 2 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 4 | 0
Nausea (Gastrointestinal disorders) | 14 | 9 | 7 | 7 | 0
Constipation (Gastrointestinal disorders) | 12 | 7 | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 8 | 5 | 6 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 2 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0
Fatigue (General disorders) | 21 | 14 | 14 | 6 | 2
Gait disturbance (General disorders) | 3 | 0 | 4 | 3 | 0
Oedema peripheral (General disorders) | 2 | 0 | 4 | 2 | 2
COVID-19 (Infections and infestations) | 3 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 4 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 10 | 5 | 1 | 4 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 3 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 4 | 2 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 10 | 5 | 1 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 5 | 1 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
Seizure (Nervous system disorders) | 6 | 3 | 3 | 2 | 0
Hemiparesis (Nervous system disorders) | 2 | 3 | 5 | 3 | 0
Headache (Nervous system disorders) | 6 | 5 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 2 | 2 | 2 | 0
Facial paresis (Nervous system disorders) | 3 | 0 | 1 | 2 | 1
Aphasia (Nervous system disorders) | 3 | 3 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 2 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 2 | 0
Memory impairment (Nervous system disorders) | 3 | 2 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 3 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 5 | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 1 | 0 | 2 | 0
Agitation (Psychiatric disorders) | 2 | 2 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 3 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 4 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 5 | 2 | 2 | 1 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated during the Phase 1b portion of the trial as the initial responses to selinexor treatment were not supportive of continued investigation in glioblastoma, therefore there was no reporting of the Phase 2 outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT04421378/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT04421378/SAP_001.pdf